CLINICAL TRIAL: NCT04911556
Title: Study for the Effect of Probiotics on Aging Population
Brief Title: the Effect of Probiotics on Aging Population
Acronym: TEOPOGP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wuxi People's Hospital (Other)
Collaborators: Jiangnan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z202002
Record Dates: First submitted 2021-05-12; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Debility
Keywords: intestinal flora
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: One group served as a control group, while the other three groups are treated with different strains of bifidobacterium longum
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant ,care provider,investigator and outcomes Assessor are all blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- the placebo group (Placebo Comparator): A placebo made of starch
  Interventions: Dietary Supplement: A placebo made of starch
- Bifidobacterium longum group 1 (Experimental): Bifidobacterium longum 274
  Interventions: Dietary Supplement: Bifidobacterium longum
- Bifidobacterium longum group 2 (Experimental): Bifidobacterium longum 4-1
  Interventions: Dietary Supplement: Bifidobacterium longum
- Bifidobacterium longum group 3 (Experimental): Bifidobacterium longum gs
  Interventions: Dietary Supplement: Bifidobacterium longum

INTERVENTIONS:
Dietary Supplement: Bifidobacterium longum — types of intestinal flora
  Arms: Bifidobacterium longum group 1; Bifidobacterium longum group 2; Bifidobacterium longum group 3
Dietary Supplement: A placebo made of starch — placebo
  Arms: the placebo group

SUMMARY:
This study intends to recruit aging population (over 65 years old). The investigators use 16 SrDNA sequencing technology, genome sequencing technology, metabonomics, random forest forecast model, analysing and selecting specific age-related intestinal flora. The investigators select probiotics slowing down senility. Then the investigators use the probiotics to intervene in the aging population. Finally the investigators observe whether the probiotics can delay aging.

DETAILED DESCRIPTION:
This project plans to recruit the aging population (aged over 65 years old) and comprehensively analyze the public database and self-sequencing clinical big data by using 16 srDNA sequencing technology, metagenomic sequencing technology, metabonomics methods and Random Forest (R) prediction model to judge the key bacterial communities and related functional pathways related to aging.Based on the analysis results, the probiotics with the potential to alleviate aging were selected for intervention evaluation of aging population. This topic aims to explore the change process of intestinal flora structure and composition related to aging process.Identify the key intestinal bacteria genera/species/strains associated with aging, and target the pathway and metabolic characteristic spectrum of the key bacterial communities associated with aging;And select and breed specific intestinal bacterial strains related to aging.The aim is to reduce the age-related metabolic abnormalities and chronic inflammation, reduce medical treatment, rationally allocate medical resources, reduce medical costs and improve the quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Over 65 years old
2. Frail scale score above 3 points

Exclusion Criteria:

1. Severe impairment of liver and kidney function
2. The tumor is advanced and life expectancy is less than 2 years
3. Severe cognitive impairment and inability to cooperate
4. Unable to give informed consent
5. Have participated in other study before

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Points of probiotics intervention in aging population | one year
  The score of Frail scale 0 points is defined as normal.And 1 to 3 points is defined as the early age of debility.Three points or more is defined as debility.The score is lower than before, meaning probiotic intervention can alleviate debility.

CONTACTS AND LOCATIONS:
Overall Officials: Kan Hong, doctor, Study Director — Wuxi People's hospitial

IPD SHARING:
Plan to Share IPD: No